CLINICAL TRIAL: NCT04702828
Title: Fall Syndrome: The Influence Of Physiological And Psychological Factors On Behavior After Falls Principal Investigator
Brief Title: The Influence Of Physiological And Psychological Factors On Fall Syndrome
Status: Completed | Type: Observational
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Shu-Chun Lee, Principal Investigator, Taipei Medical University
Other Study IDs: N202002009
Record Dates: First submitted 2021-01-07; First posted 2021-01-11 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Fall
Keywords: Fall Syndrome, elderly,Physiological,Psychological

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fallers group: 1.60 years to 99 years old 2. have a recent fall within two months 3.can understand and answer the questions 4.can give their informed consent
- Non-fallers group: 1.60 years to 99 years old 2. have any fall experiences in past year 3.can understand and answer the question 4.can give their informed consent

SUMMARY:
Most of previous studies are cross-sectional studies, and rarely explore the changes in physical activity, mental state, cognitive and motor functions over time after a fall. Therefore, we hope to find out what changes in the elders' physiological and psychological functions after a fall.

DETAILED DESCRIPTION:
Falls are the main cause of accidental injuries that are common among the elderly. In Taiwan, the incidence of falls is about 15% to 34%. Falling can cause subsequent serious injuries and post-fall syndromes. Post-fall syndrome is common after a fall. The symptoms of self-restricted activity for fear of falling again affect about one-fifth of older fallers. This syndrome develops within a short period of time after a fall, which not only causes serious problems but also affects psychological symptoms and dependence on daily life functions. All of these reduce the function of movement and increase the chance of falling again. However, most of the past studies are cross-sectional studies, and rarely explore the changes in physical activity, mental state, cognitive and motor functions over time after a fall. Therefore, the study will investigate the changes in physiological and psychological functions after a fall among older adults who experiences a recent fall within 2 months. Additionally, the physiological and psychological functions will be compared between older adults with and without a history of falls.

ELIGIBILITY:
Inclusion Criteria:

1.60 years to 99 years old 2.Fall experiences within two months 3.Can understand and answer the questions 4.Can give their informed consent

Exclusion Criteria:

1.Serious fracture or head trauma caused by a fall, 2.Unable to perform a walking test, 3. Neurological diseases

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Older participants with a history of fall within 2 months will be recruited from the emergency department in a regional hospital and older participants without a history of fall in the past year will be recruited from the community daycare centers.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2021-03-02 (Actual); Study Completion 2021-03-02 (Actual)

PRIMARY OUTCOMES:
Visual acuity | Baseline
  Vision acuity will be measured by the Snellen Chart. The Snellen chart is printed with eleven lines of block letters. The first line consists of one very large E letter. Subsequent rows have increasing numbers of letters with decrease in size. Participant will take the test by covering one eye from 6 meters away, and read aloud the letters of each row, beginning at the top. The smallest row that can be read accurately indicates the visual acuity in that specific eye.
Vertigo symptom | Baseline
  Situational Vertigo Questionnaire (SVQ) consists of 19 questions, with a score from 0 (not at all), 1 (very slightly), 2 (somewhat), 3 (quite a lot) to 4 (very much). It measures how frequently symptoms (unusual disorientation, dizziness, giddiness, light-headedness or unsteadiness) are provoked or exacerbated in environments with visual-vestibular conflict or intense visual motion e.g. busy supermarket aisles. A score is obtained by dividing the total sum for activities experienced by the number of activities.
Medication history | Baseline
  Medication history will be recorded including drug name, dose, route, and frequency.
Static balance | Baseline
  Static balance test will be assessed by the modified Clinical Test for Sensory Interaction in Balance(mCTSIB), The mCTSIB was developed as a clinical version of the Sensory Organization Test and was developed to assess sensory contributions to postural control.
  Participants will stand with their hands at their sides, feet together and perform the following 4 sensory conditions: (1) Stand on firm surface, eyes open (2) Stand on firm surface, eyes closed (3) Stand on foam surface, eyes open (4) Stand on foam surface, eyes closed. Each condition will be timed for maximum 30 seconds. The test is terminated when a participant's arms or feet move. If a participant is unable to maintain the position for 30 seconds they are provided with 2 additional attempts. The time (s) to complete each condition will be recorded.
Dynamic balance | Baseline
  Dynamic balance test will be evaluated by the functional reach test. The participant will be instructed to stand next to a wall and position the arm that is closer to the wall at 90 degrees of shoulder flexion. The assessor instructs the participant to "Reach as far as you can forward without taking a step." The distance (cm) from the start to end position at the middle fingertip will be measured.
Walking ability | Baseline
  Walking ability test will be measured by the 10 meter walk test. Participant will be asked to walk on a 14 meters walkway at their comfortable speed. The time for the middle 10 meters will be recorded and walking speed (m/s) will be calculated.
Hand grip | Baseline
  Dominant hand grip (kg) will measured by a dynamometer. Participants will stand with their arms down by their sides. They will squeeze the dynamometer with maximum isometric effort, which is maintained for 6 seconds.
Lower limbs strength | Baseline
  Lower limbs strength will be assessed by the Five Times Sit to Stand. Participants will be asked to sit on the chair with arms folded across their chest, and stand up and sit down as quickly as possible for 5 times. The time (s) to complete the task will be recorded.
Function ability | Baseline
  Function ability test will be determined by the timed up and go test (TUG). Participants will be asked to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down. The time (s) to complete the task will be recorded.
Cognitive function (mild cognitive impairment) | Baseline
  Cognitive function will be evaluated by the Montreal Cognitive Assessment (MoCA), which covers visuospatial abilities, short-term memory recall task, multiple aspects of executive functions, attention, concentration, and working memory. The total score is 30 and cut-off point is 26. Score less than 26 indicates mild cognitive impairment.
Cognitive function (dementia) | Baseline
  Mini-Mental State Examination(MMSE) is used extensively in clinical and research settings to measure cognitive impairment, covering attention, calculation, recall, language, ability to follow simple commands and orientation. It is commonly used in medicine and allied health to screen for dementia; used to estimate the severity and progression of cognitive impairment and to follow the course of cognitive changes in an individual over time; thus making it an effective way to document an individual's response to treatment.
Fear of falling | Baseline
  Fear of falling will be measured by the Falls Efficacy Scale International(FES). The FES rated each daily task from no confident at all to completely confident. The total score between 16 and 64, and the score more than 28 indicates higher level of fear of falling.
The confidence of balance | Baseline
  The confidence of balance will test by Activities-specific Balance and Confidence (ABC) Scale. The ABC Scale is a 16-item questionnaire. Each item is rated from 0% (no confidence) to 100% (complete confidence) by all participants. The higher score, the more confidence they have.
Depression Anxiety and Stress | Baseline
  Depression, anxiety and stress will be assessed by the Depression Anxiety and Stress(DASS-21). It is a self-reported scale designed to measure the negative emotional states of depression, anxiety and stress. The higher score indicates the increased severity of symptoms.
Sarcopenia | Baseline
  Sarcopenia will be screened by the SARC-F including how much difficulty do you have in lifting and carrying 10 pounds, how much difficulty do you have walking cross a room, how much difficulty do you have transferring from a chair or bed, how much difficulty do you have climbing a flight of 10 stairs, and how many times have you fallen in the past year. The score more than 4 indicates high risk of sarcopenia.
Frailty | Baseline
  Frailty will be assessed by the Fried frailty phenotype. It is a yes-no model based on five items including physical inactivity, low muscle strength, slow gait speed, exhaustion/ fatigue and weight loss. Each item is scored as 0 (no) or 1 (yes). The score of greater than 3 indicates frailty.
Basic Activity of Daily Living | Baseline
  Basic activities of daily living will be measured by the Barthel Index. It is an ordinal scale used to measure performance in activities of daily living (ADL). Ten variables describing ADL and mobility are scored, a higher number being a reflection of greater ability to function independently following hospital discharge. Time taken and physical assistance required to perform each item are used in determining the assigned value of each item. The Barthel Index measures the degree of assistance required by an individual on 10 items of mobility and self care ADL. The score of 0-20 indicates "total" dependency, 21-60 indicates "severe" dependency, 61-90 indicates "moderate" dependency, and 91-99 indicates "slight" dependency.
Instrumental Activity of Daily Living | Baseline
  Instrumental activities of daily living (IADL) will be measured by the Lawton Instrumental Activities of Daily Living Scale which assesses a person's ability to perform tasks such as using a telephone, doing laundry, and handling finances. It contains eight items, with a summary score from 0 (low function) to 8 (high function).
Health-related quality of life | Baseline
  The quality of life will be assessed by the Control, Autonomy, Self-Realization and Pleasure (CASP-19), which has 4 subscales and 19 items in total. A 4-point Likert scale is used including "often", "sometimes", "not often" and "never". The higher score indicates the better quality of life.
Physical Activity | Baseline
  Physical Activity will be examined by the International Physical Activity Questionnaire (IPAQ)-Short Form. Participants will be asked about their duration (in minutes) and frequency (days) when performing four specific types of activity: walking, moderate intensity, vigorous intensity and sitting.
Social function survey | Baseline
  Participants will be asked whether they have been in contact with family or friends in the past six months. According to the scale of different networks, the frequency of interaction and the degree of closeness, interpersonal relationships and social support networks can be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Chun Lee, PhD, Principal Investigator — School of Gerontology Health Management
Locations (1):
- Community Daycare Center, Taipei, Taiwan